CLINICAL TRIAL: NCT07066488
Title: Brief Group Intervention Based on Acceptance and Commitment Therapy (ACT) for Problem Gambling: A Pilot Study
Brief Title: Brief ACT Intervention for Problem Gambling: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-81
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Problem Gambling
Keywords: Problem Gambling; Gaming Disorder; Psychological Inflexibility
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT group (Experimental): 8 group weekly sessions including ACT methods
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Acceptance and Commitment Therapy methods were focused on promoting Values clarification, Acceptance, Cognitive defusion, Committed action and Flexible attention to the present moment, and included methods such as the Garden Metaphor or defusion training.

SUMMARY:
The goal of this pilot study is to learn if Acceptance and Commitment Therapy (ACT) works to treat Problem Gambling in young adults.The main questions it aims to answer are:

* Does ACT therapy improve health and gambling behavior?
* Is an 8-week online group therapy format viable for youth with gambling problems? Researchers will assess whether changes in health, gambling behavior, and other psychological variables are observed after eight weeks of therapy.

Participants will:

* Attend weekly online group sessions for 8 weeks
* Learn new tools that they will put into practice after the sessions
* Be required to complete evaluation questionnaires before and after the intervention and at the 3- and 6-month follow-up

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will be assessed to determine eligibility for study entry.

Patients who meet eligibility requirements will receive psychological intervention consisting in an 8-session group on line-delivered ACT-based treatment.

The participants will be assessed through self-report instruments before and after treatment and at 3 and 6 months follow-up.

The pilot study will not include a control group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years
* Score ≥ 3 on the Problem Gambling Severity Index (PGSI)
* Comprehension of Spanish, online connection, and signed consent

Exclusion Criteria:

* In active psychological or pharmacological treatment for gambling disorder
* Having received ACT-based psychological treatment in the last 6 months
* Problematic substance use: CAGE Adapted to Include Drugs Questionnaire (CAGE-AID) score ≥ 3
* Difficulty consistently attending online sessions

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Problem Gambling Severity Index (PGSI) | Change from Baseline severity of problem gambling at 8 months
  The PGSI is a 9-item, 4-point Likert-format self-report scale (0 = never, 3 = almost always) that assesses the severity of problem gambling. Scores range from 0 to 27. A score of 8 or higher is considered indicative of problem gambling. Higher scores indicate greater severity of the disorder.

SECONDARY OUTCOMES:
Change in Difficulties in Emotion Regulation Scale (DERS-28) | Change from Baseline emotion regulation at 8 months
  The DERS-28 is a 28-item questionnaire with a 5-point Likert format (1 = almost never, 5 = almost always) that assesses difficulties in emotion regulation. It consists of six subscales: emotional nonacceptance, difficulty achieving goals, impulsivity, emotional awareness, limited strategies, and emotional clarity. Higher scores indicate greater difficulties in emotional regulation and worse clinical outcomes.
Change in General Health Questionnaire (GHQ-12) | Change from Baseline psychological distress and perceived general health at 8 months
  The GHQ-12 is a 12-item self-report questionnaire designed to detect general psychological symptoms. It is answered on a 4-point Likert-type scale. Higher scores reflect greater psychological distress and poorer perceived general health.
Change in the Comprehensive ACT Process Assessment Questionnaire (CompACT) | Change from Baseline psychological flexibility at 8 months
  The CompACT is a 23-item, 7-point Likert-format scale (0 = not at all true, 6 = completely true) that assesses psychological flexibility, a core process of Acceptance and Commitment Therapy. It includes three subscales: openness to experience, awareness, and committed action. Higher scores reflect greater psychological flexibility.
Change in Values Living Questionnaire (VLQ) | Change from Baseline value-behavior alignment at 8 months
  The Valued Living Questionnaire assesses the degree of perceived importance and consistency of action directed toward personal values in 10 life domains (family, work, health, leisure, etc.). Each item is scored from 1 to 10. A composite index of discrepancy between importance and action is calculated. Higher scores indicate less value-behavior alignment.
Change in Gambling-Related Emotional Distress Scale | Change from Baseline gambling-related distress at 8 months
  A weekly subjective scale assessing the frequency and intensity of emotional distress associated with gambling behavior using Likert scales ranging from 0 to 5. Higher scores reflect greater gambling-related distress.
Change in Gambling-Related Experiential Avoidance scale | Change from Baseline Experiential Avoidance at 8 months
  A weekly subjective scale assessing the extent to which the participant has attempted to avoid gambling-related emotions, thoughts, or internal situations. Higher scores indicate greater experiential avoidance and less flexibility.
Change in the frequency of self-reported gambling behaviors | Change from Baseline gambling behaviors at 8 months
  Daily self-monitoring in which the participant indicates whether they gambled, the duration, type of gambling, emotions before, during, and after, and perceived function of the behavior. Weekly frequency of gambling episodes will be analyzed. Higher frequency is interpreted as worse clinical outcome.
Change in the frequency of committed actions | Change from Baseline committed actions at 8 months
  Self-monitoring of the frequency with which the participant has acted in accordance with their personal values during moments of desire to gamble. This is considered a positive behavioral indicator of change.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Montesinos, Ph.D., Principal Investigator — Universidad Europea de Madrid; David Lobato, Ph.D., Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT07066488/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT07066488/ICF_001.pdf